CLINICAL TRIAL: NCT04679038
Title: SHR-1701 Plus Famitinib Malate in Advanced Solid Tumors: An Open-label, Multi-center, Phase I/II Trial
Brief Title: A Trial of SHR-1701 in Combination With Famitinib in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1701-II-203
Record Dates: First submitted 2020-12-14; First posted 2020-12-22 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Solid Tumor
MeSH Terms: interventions — SHR-1701; famitinib

STUDY DESIGN:
Intervention Model Description: SHR-1701 plus famitinib
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combinational therapy part (Experimental): SHR-1701 + famitinib
  Interventions: Biological: SHR-1701; Drug: Famitinib
- monotherapy part (Experimental): famitinib
  Interventions: Drug: Famitinib

INTERVENTIONS:
Biological: SHR-1701 — Intravenous (IV) on Day 1 of each cycle
  Arms: combinational therapy part
Drug: Famitinib — Famitinib, po, qd

SUMMARY:
This is an open-label, multi-center study to evaluate the efficacy and safety of SHR-1701 in combination with famitinib in subjects with metastatic or locally advanced solid tumor. There are two parts of the study: combinational therapy part and monotherapy part. Phase I of combinational therapy part is to determine the recommended dose for Phase II (RP2D) for famitinib in the combined regimen, then efficacy and safety of SHR-1701 plus famitinib (RP2D) will be further evaluated in the following Phase II in cohorts 1/2/3, with simon's two-stage design. Meanwhile, efficacy and safety of famitinib will also be assessed in cohorts 4/5 in the monotherapy part.

ELIGIBILITY:
Inclusion Criteria:

1. Phase I of combinational therapy part: Histologically proven metastatic or locally advanced solid tumors, for which no effective standard treatment exists or standard therapy has failed.
2. Phase II of combinational therapy part and monotherapy part: Histologically confirmed metastatic or locally advanced selected solid tumor types with 0-2 prior lines of systemic therapy.

   For cohorts 1 or 4, patients with biliary tract carcinoma failed to one prior systemic treatment. Patients with previous adjuvant/neo-adjuvant therapy completed within 6 months can be enrolled.

   For cohort 2, patients with clear-cell renal cell carcinoma (or predominantly clear-cell subtype with primary tumor resected) after failure of no more than first-line standard therapy; For cohorts 3 or 5, patients with hepatocellular carcinoma must have progressed on prior first- or second-line standard therapy; Child-Pugh Class A; BCLC stage B or C, and not suitable for surgical or local therapy.
3. Subjects are 18 years old or older when signing the informed consent and gender is not limited.
4. Life expectancy of at least 12 weeks.
5. Eastern Cooperative Group (ECOG) performance status of 0 to 1.
6. At least one measurable lesion according to RECIST version 1.1.
7. Tumor tissue must be available for biomarker analysis prior to the first dose of treatment, If not available, subjects can consult the investigator for enrollment agreement.
8. Adequate hematological, hepatic and renal function as defined in the protocol.
9. Subjects with HBV infection: HBV DNA<500 IU/mL or < 2500 copy/mL, must receive anti-HBV therapy.
10. Subjects with HCV-RNA(+) must receive antiviral therapy.
11. Able and willing to provide signed informed consent form, and able to comply with all procedures.

Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

1. For cohorts 1 or 4: known ampullary cancer or mixed cancer (HCC-ICC).
2. For cohorts 3 or 5: known hepatocholangiocarcinoma, sarcomatoid HCC, mixed cell carcinoma and lamellar cell carcinoma; history of hepatic encephalopathy.
3. For subjects in combinational therapy part: prior treatment with any anti-PD-1/PD-L1, or anti-CTLA-4 agents (specifically targeting T-cell co-stimulation or checkpoint pathways), or TGF-β inhibitors.
4. For cohort 4: prior treatment with VEGFR directed therapies including famitinib.
5. Factors to affect oral administration.
6. Major surgery procedure within 28 days prior to the first dose of trial treatment (excluding prior diagnostic biopsy or PICC); anticancer treatment within 28 days before the first dose of trial treatment; subjects in combinational therapy part who have received systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to the first dose of trial treatment should also be excluded.
7. Moderate-to-severe ascites with clinical symptoms.
8. Active or history of central nervous system metastases.
9. Known genetic or acquired hemorrhage or thrombotic tendency.
10. History of gastrointestinal hemorrhage within 6 months prior to the start of study treatment or clear tendency of gastrointestinal haemorrhage.

Other protocol defined exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
RP2D | First cycle (21 days)
  Recommended phase-2 dosage
Objective response rate (ORR) | up to approximately 3 years (anticipated)
  Defined as complete or partial response per RECIST 1.1

SECONDARY OUTCOMES:
Clinically Significant Toxicity | First cycle (21 days)
  Number of subjects in Phase I of combinational therapy part who experienced clinically significant toxicity
AEs+SAEs | up to approximately 3 years (anticipated)
  The incidence and severity of Adverse Events and Serious Adverse Events
DCR | up to approximately 3 years (anticipated)
  Disease Control Rate per RECIST 1.1
DoR | up to approximately 3 years (anticipated)
  Duration of Response per RECIST 1.1
PFS | up to approximately 3 years (anticipated)
  Progression-Free-Survival
OS | up to approximately 3 years (anticipated)
  OS is the time interval from the start of treatment to death from any cause or lost of follow-up
6-month OS rate | From the start of treatment to 6 months
  6-month-overall survival rate
12-month-OS rate | From the start of treatment to 12 months
  12-month- overall survival rate
Cmax of SHR-1701 | up to approximately 3 years (anticipated)
  Maximum Plasma Concentration of SHR-1701
C6h of Famitinib | up to approximately 6 months (anticipated)
  Plasma Concentration of 6 hours after famitinb administration
Cmax,ss | up to approximately 3 years (anticipated)
AUC0-24h,ss | up to approximately 3 years (anticipated)]

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The 2nd Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Gannan, Jiangxi
  - Jinan Central Hospital, Jinan, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - Huashan Hospital,Fudan University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - The 2nd Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The 1st Affiliated Hospital of Zhejiang Medical University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No